CLINICAL TRIAL: NCT00659659
Title: A Phase 1, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Effects of MEDI-563, A Humanized Anti-Interleukin-5 Receptor Alpha Monoclonal Antibody, on Airway Eosinophils in Adults With Atopic Asthma
Brief Title: A Study to Evaluate the Safety, Tolerability and Effects of MEDI-563 in Adults With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP166
Record Dates: First submitted 2008-04-11; First posted 2008-04-16 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): MEDI-563
  Interventions: Drug: MEDI-563
- 2 (Experimental): MEDI-563
  Interventions: Drug: MEDI-563
- 4 (Placebo Comparator): Placebo
  Interventions: Other: Placebo Comp.
- 5 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MEDI-563 — 1.0 mg/kg IV: MEDI-563
  Arms: 1
Drug: MEDI-563 — 100 mg, 200 mg SC
  Arms: 2
Other: Placebo Comp. — Placebo SC
  Arms: 4
Other: Placebo — Placebo as a single IV infusion (Certain number of subjects)
  Arms: 5

SUMMARY:
Evaluate the safety and tolerability of MEDI-563 in adults with asthma and the effects of MEDI-563 on eosinophil counts in airway mucosal biopsies

DETAILED DESCRIPTION:
Evaluate the safety and tolerability of MEDI-563 in adults with atopic asthma; and evaluate the effects of MEDI-563 on eosinophil counts in airway mucosal biopsies 28 days after completion of dosing in adults with atopic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults, 18 through 65 years of age at time of randomization;
* Written informed consent obtained from the subject prior to beginning study procedures or receipt of any study medication;
* Previously documented diagnosis of asthma of ≥ 1 year duration, based on episodic symptoms of airflow obstruction; post-bronchodilator reversibility of airflow obstruction ≥ 12% (in USA only - if subject does not achieve this during screening, proof of ≥12% reversibility within 1 year of randomization is acceptable) or proof of a positive response to a methacholine challenge during screening with prior approval from MedImmune (in USA only - within 1 year of randomization is acceptable) as represented by a provoking concentration of methacholine to cause a 20% fall in FEV1 (PC20) < 8 mg/ml [American Thoracic Society (ATS), 2000)]; and exclusion of alternative pulmonary diagnoses (eg, cystic fibrosis, COPD);
* Asthma symptoms are adequately controlled on a therapeutic regimen that has not changed in the last 4 weeks prior to Study Day 0, and the subject is willing to maintain the same therapeutic regimen and doses from the time of screening to the time of the first follow-up bronchoscopy with airway mucosal biopsies (Study Day 28 for Cohort 1; Study Day 84 for Cohort 2);
* Pre-bronchodilator FEV1/forced vital capacity (FVC) ratio that is below the age-adjusted normal limit as defined by the 2007 National Heart Lung and Blood Institute Asthma guidelines (Appendix D) and post-bronchodilator FEV1 ≥ 65% at screening;
* Must have ≥ 2.5% eosinophils in sputum;
* Have had no hospitalizations due to asthma in the last year prior to screening;
* Women of childbearing potential, unless surgically sterile or at least 1 year post-menopausal, must use 2 effective methods of avoiding pregnancy
* Able to complete the follow-up period as required by the protocol;
* Willing to forego other forms of experimental treatment and study procedures during the study and during an 84-day period after the last dose of study drug;
* Able to provide spirometric readings that meet ATS standards

Exclusion Criteria:

* Participation in any previous MEDI-563 clinical study;
* Known history of allergy or adverse reactions to any component of the study drug formulation;
* Lung disease other than asthma (eg, COPD, cystic fibrosis, eosinophilic pneumonia);
* Current use of any systemic or inhaled immunosuppressive drugs [oral (up to a maximum dose of 10 mg/day or 20 mg every other day) and inhaled corticosteroids are allowed if dose has been stable for at least 4 weeks prior to study drug administration on Study Day 0].
* Current use of any β-blocker (eg, propranolol);
* Acute illnesses or evidence of clinically significant active infection, such as fever ≥ 38.0ºC (100.5ºF) at screening and through the time of the study drug administration on Study Day 0;
* Receipt of any investigational drug therapy, intravenous immunoglobulin (IVIG), or monoclonal therapy (eg, Xolair) within 30 days or within 5-half lives prior to study drug administration on Study Day 0 through End of Study/Study Termination (Study Day 84 for Cohort 1 or Study Day 140 for Cohort 2);
* Pregnancy (women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to study drug administration on Study Day 0);
* Breastfeeding or lactating;
* History of alcohol or drug abuse < 1 year prior to Study Day 0;
* History of cancer, apart from basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy > 1 year prior to Study Day 0;
* History of a previous episode of active TB or a positive TB skin test without completion of an appropriate course of treatment;
* A history of coagulation disorders that would contraindicate mucosal biopsies;
* History of immunodeficiency or infection with HIV-1, HIV-2, or hepatitis A, B, or C virus;
* History of use of tobacco products within 2 years of baseline (Study Day 0) or history of smoking ≥ 10 pack-years;
* Elective surgery planned from the time of screening through first follow-up bronchoscopy with airway mucosal biopsies (Study Day 28 or Study Day 84, as applicable);
* Evidence of any systemic disease or respiratory disease (other than asthma), history of any disease, or any finding upon physical examination, screening laboratory test, chest X-ray (CXR), or ECG that, in the opinion of the investigator or medical monitor, may compromise the safety of the subject in the study or confound the analysis of the study results;
* Any employee of the research site who is involved with the conduct of the study;
* History of lidocaine allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of MEDI-563 in adults with atopic asthma and evaluate the effects of MEDI-563 on eosinophil counts in airway mucosal biopsies 28 days after completion of dosing in adults with atopic asthma. | Study Day 84 or Day 140 - (dose-driven)

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics (PK) of MEDI-563 in adults with atopic asthma, and evaluate the immunogenicity (IM) of MEDI-563 in adults with atopic asthma. | Day 84 or 140

CONTACTS AND LOCATIONS:
Overall Officials: David Gossage, M.D., MBA, Study Director — MedImmune LLC
Locations (10):
- United States (5):
  - Research Site, Denver, Colorado
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, Madison, Wisconsin
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec

REFERENCES:
- [Derived] Chachi L, Diver S, Kaul H, Rebelatto MC, Boutrin A, Nisa P, Newbold P, Brightling C. Computational modelling prediction and clinical validation of impact of benralizumab on airway smooth muscle mass in asthma. Eur Respir J. 2019 Nov 14;54(5):1900930. doi: 10.1183/13993003.00930-2019. Print 2019 Nov. No abstract available. PMID 31391226